CLINICAL TRIAL: NCT01055314
Title: A Pilot Study to Evaluate Novel Agents (Temozolomide and Cixutumumab [IMC-A12, Anti-IGF-IR Monoclonal Antibody NSC # 742460]) in Combination With Intensive Multi-agent Interval Compressed Therapy for Patients With High-Risk Rhabdomyosarcoma
Brief Title: Temozolomide, Cixutumumab, and Combination Chemotherapy in Treating Patients With Metastatic Rhabdomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02005; NCI-2011-02005 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ARST08P1; ARST08P1 (Other: Children's Oncology Group); ARST08P1 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-07

CONDITIONS: Adult Rhabdomyosarcoma; Childhood Alveolar Rhabdomyosarcoma; Childhood Embryonal Rhabdomyosarcoma; Metastatic Childhood Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma; Untreated Childhood Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma | interventions — cixutumumab; Cyclophosphamide; Dactinomycin; Doxorubicin; Etoposide; Ifosfamide; Irinotecan; Temozolomide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (chemotherapy, radiation therapy, cixutumumab) (Experimental): Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1-5, 7, 8, 11, 12, 15, 16, 20-24, 28, 29, 32, 33, 35, 38, 41-44, 47, 48, 50, and 51; irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 1, 4, 20, 23, 47, and 50; ifosfamide IV over 1 hour and etoposide IV over 1-2 hours on days 1-5 of weeks 9, 13, 17, 26, and 30; doxorubicin hydrochloride IV over 1-15 minutes on days 1 and 2 of weeks 7, 11, 15, 28, and 32; cyclophosphamide IV over 30-60 minutes on day 1 of weeks 7, 11, 15, 28, 32, 35, 38, 41, and 44; dactinomycin IV over 1-5 minutes on day 1 of weeks 35, 38, 41, and 44; and cixutumumab IV over 1 hour on day 1 of weeks 1-51. Patients also undergo radiation therapy on days 1-5 of weeks 20-24.
  Interventions: Biological: Cixutumumab; Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Ifosfamide; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Vincristine Sulfate Liposome
- Group 2 (chemotherapy, radiation therapy, temozolomide) (Experimental): Patients receive vincristine sulfate, irinotecan hydrochloride, ifosfamide, etoposide, doxorubicin hydrochloride, cyclophosphamide, and dactinomycin and undergo radiation therapy as in group 1. Patients also receive temozolomide PO on days 1-5 of weeks 1, 4, 20, 23, 47, and 50.
  Interventions: Drug: Cyclophosphamide; Biological: Dactinomycin; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Ifosfamide; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Temozolomide; Drug: Vincristine Sulfate Liposome

INTERVENTIONS:
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
  Arms: Group 1 (chemotherapy, radiation therapy, cixutumumab)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; ACTINOMYCIN D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; U-101440E
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temodal; Temodar
  Arms: Group 2 (chemotherapy, radiation therapy, temozolomide)
Drug: Vincristine Sulfate Liposome — Given IV
  Other Names: Marqibo

SUMMARY:
This randomized pilot clinical trial is studying the side effects and how well giving temozolomide and cixutumumab together with combination chemotherapy works in treating patients with metastatic rhabdomyosarcoma. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving temozolomide and cixutumumab together with combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of administering IMC-A12 (cixutumumab) in combination with a multi-agent intensive chemotherapy regimen for the treatment of high-risk rhabdomyosarcoma (RMS).

II. To determine the feasibility of adding temozolomide to vincristine (vincristine sulfate)/irinotecan (irinotecan hydrochloride) cycles in patients with high-risk RMS.

III. To assess immediate and short-term side effects of delivery of concurrent temozolomide-vincristine-irinotecan with irradiation in patients with high-risk RMS.

SECONDARY OBJECTIVES:

I. To gain a preliminary estimate of the response rate to IMC-A12 or temozolomide plus vincristine/irinotecan in previously untreated high-risk RMS.

II. To obtain preliminary efficacy data for IMC-A12 or temozolomide in combination with a multi-agent interval compressed chemotherapy regimen in previously untreated high-risk RMS.

III. To determine the effectiveness of detecting metastatic disease with fludeoxyglucose F 18 positron emission tomography (FDG PET) and to compare assessment of response using standard imaging techniques with response assessed by FDG PET.

IV. To assess changes in serum levels of insulin-like growth factor (IGF)-I, IGF-II, IGF-BP3 as biomarkers of IGF-IR inhibition.

OUTLINE: This is a dose-escalation study of cixutumumab. Patients are assigned to 1 of 2 treatment groups according to the timing of their enrollment onto the study.

GROUP 1: Patients receive vincristine sulfate intravenously (IV) over 1 minute on day 1 of weeks 1-5, 7, 8, 11, 12, 15, 16, 20-24, 28, 29, 32, 33, 35, 38, 41-44, 47, 48, 50, and 51; irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 1, 4, 20, 23, 47, and 50; ifosfamide IV over 1 hour and etoposide IV over 1-2 hours on days 1-5 of weeks 9, 13, 17, 26, and 30; doxorubicin hydrochloride IV over 1-15 minutes on days 1 and 2 of weeks 7, 11, 15, 28, and 32; cyclophosphamide IV over 30-60 minutes on day 1 of weeks 7, 11, 15, 28, 32, 35, 38, 41, and 44; dactinomycin IV over 1-5 minutes on day 1 of weeks 35, 38, 41, and 44; and cixutumumab IV over 1 hour on day 1 of weeks 1-51. Patients also undergo radiation therapy* on days 1-5 of weeks 20-24.

GROUP 2: Patients receive vincristine sulfate, irinotecan hydrochloride, ifosfamide, etoposide, doxorubicin hydrochloride, cyclophosphamide, and dactinomycin and undergo radiation therapy* as in group 1. Patients also receive temozolomide orally (PO) on days 1-5 of weeks 1, 4, 20, 23, 47, and 50.

GROUP 3: Patients receive vincristine sulfate, irinotecan hydrochloride, ifosfamide, etoposide, doxorubicin hydrochloride, cyclophosphamide, dactinomycin, and cixutumumab and undergo radiation therapy* as in group 1. Patients also receive temozolomide as in group 2. (Discontinued as of January 2013)

NOTE: *Patients with parameningeal tumors and evidence of intracranial extension or those requiring emergency radiotherapy may receive radiation therapy starting in week 1; cixutumumab should be withheld during radiation therapy.

After completion of study therapy, patients are followed up at 3 weeks and then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be eligible for, and enrolled on D9902 prior to enrollment on ARST08P1
* Patients with newly diagnosed, biopsy-proven metastatic rhabdomyosarcoma or ectomesenchymoma (stage IV, clinical group IV) are eligible for this study; patients with stage IV, clinical group IV RMS with parameningeal and paraspinal primary tumors, including those with intracranial extension (ICE) are eligible for ARST08P1; ICE is defined by contrast magnetic resonance imaging (MRI) showing that the primary tumor touches, displaces, invades, distorts, or otherwise causes signal abnormality of the dura in brain or spinal cord in contiguity to the primary site; ICE is also presumed to exist if the cerebrospinal fluid (CSF) cytopathology is positive for tumor at diagnosis
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* No prior chemotherapy or radiotherapy except for use of corticosteroids or emergent radiation therapy; patients requiring emergency radiation are eligible
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73m^2 OR maximum serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (for patients 1 to 5 months of age)
  * 0.5 mg/dL (for patients 6 to 11 months of age)
  * 0.6 mg/dL (for patients 1 year of age)
  * 0.8 mg/dL (for patients 2 to 5 years of age)
  * 1.0 mg/dL (for patients 6 to 9 years of age)
  * 1.2 mg/dL (for patients 10 to 12 years of age)
  * 1.5 mg/dL (males) or 1.4 mg/dL (females) (for patients 13 to 15 years of age)
  * 1.7 mg/dL (males) or 1.4 mg/dL (females) (for patients >= 16 years of age)
* Patients with urinary tract obstruction by tumor must meet the renal function criteria listed above AND must have unimpeded urinary flow established via decompression of the obstructed portion of the urinary tract
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age, unless there is evidence of biliary obstruction by the tumor
* Shortening fraction >= 27% by echocardiogram (ECHO) OR ejection fraction >= 50% by radionuclide angiogram
* Absolute neutrophil count (ANC) >= 750/uL; abnormal blood counts are permissible if there is bone marrow biopsy or aspirate proven bone marrow involvement by rhabdomyosarcoma
* Platelet count >= 75,000/uL; abnormal blood counts are permissible if there is bone marrow biopsy or aspirate proven bone marrow involvement by rhabdomyosarcoma
* Sexually active patients of childbearing potential must agree to use effective contraception during therapy (Pilots 1 and 2) and for at least 3 months after the last dose of IMC-A12 (Pilots 1)

Exclusion Criteria:

* Female patients who are pregnant are not eligible
* Female patients who are breastfeeding are not eligible; female patients who are lactating must agree to stop breastfeeding to participate in this study
* Patients receiving growth hormone therapy are not eligible
* Patients with known type I or type II diabetes mellitus are not eligible for enrollment on Pilot 1
* Patients with evidence of uncontrolled infection are not eligible
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2010-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Malempati, MD, Principal Investigator — Children's Oncology Group
Locations (139):
- United States (121):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Healthcare System - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - New York University Langone Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont College of Medicine, Burlington, Vermont
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- Starship Children's Hospital, Grafton, Auckland, New Zealand

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants started is 175. Eight patients were declared ineligible by the study chair, and one patient didn't receive treatment.
Groups:
- IMC-A12: IMC-A12 + Multi-agent intensive chemotherapy regimen.
- Temozolomide: Add temozolomide to vincristine/irinotecan cycles.
Period: Overall Study
Arm/Group | IMC-A12 | Temozolomide
Started | 100 | 75
Completed | 55 | 37
Not Completed | 45 | 38
Not completed — Adverse Event | 7 | 4
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 11 | 19
Not completed — Physician Decision | 10 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible | 3 | 5
Not completed — Refusal of further protocol therapy | 10 | 4
Not completed — No treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: 175 patients were enrolled on the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMC-A12 | Temozolomide | Total
Number analyzed (Participants) | 100 | 75 | 175
Age, Continuous [Mean (Standard Deviation); unit: Months] | 161.93 (67.36) | 152.04 (79.20) | 157.69 (72.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 30 | 83
  Male | 47 | 45 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 18 | 35
  Not Hispanic or Latino | 77 | 55 | 132
  Unknown or Not Reported | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 12 | 10 | 22
  White | 74 | 53 | 127
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Addition of Cixutumumab to Chemotherapy Determined by Patient Enrollment
Description: Proportion of no Grade 3+ cardiac toxicity.
Time Frame: From start to week 26 of therapy
Population: 18 participants were excluded because of ineligibility or insufficient information to assess feasibility.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | IMC-A12
Number analyzed (Participants) | 82
Proportion of Participants | 0.9390 [0.8872 to 0.9908]

2. Primary Outcome: Feasibility of the Addition of Temozolomide to Chemotherapy Determined by Patient Enrollment
Description: Proportion of no Grade 4+ non-hematologic toxicity.
Time Frame: From start to week 26 of therapy
Population: 13 participants were excluded because of ineligibility or insufficient information to assess feasibility.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 62
Proportion of Participants | 0.7097 [0.5967 to 0.8227]

3. Primary Outcome: Incidence of Adverse Events Assessed by Common Terminology Criteria for Adverse Events Version 4.0
Description: Number of patients with grade 3+ adverse events (AE) during therapy. (Grade 3+) = (Grade 3 + Grade 4 + Grade 5) . Grade 3: Severe and undesirable AE; Grade 4: Life threatening or disabling AE; Grade 5: Death related to AE.
Time Frame: Up to 54 weeks
Population: 9 participants who were ineligible or did not receive treatment were excluded.
Measure: Number; unit: Participants
Arm/Group | IMC-A12 | Temozolomide
Number analyzed (Participants) | 96 | 70
Participants | 89 | 61

4. Primary Outcome: Event-Free Survival
Description: Probability of no relapse, secondary malignancy, or death after 3 years in the study.
Time Frame: 3 years
Population: 9 participants who were ineligible or did not receive treatment were excluded.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | IMC-A12 | Temozolomide
Number analyzed (Participants) | 96 | 70
Probability | 0.1627 [0.0747 to 0.2507] | 0.1919 [0.0407 to 0.3431]

5. Secondary Outcome: Response Rate (CR + PR)
Description: Proportion of patients with complete or partial response. Complete Response (CR): Complete disappearance of the tumor confirmed at > 4 weeks. Partial Response (PR): At least 64% decrease in volume compared to the measurement obtained at study enrollment; Overall Response (OR) = CR + PR.
Time Frame: From the start of treatment until a maximum of 2 cycles (21 days per cycle) of treatment in the absence of disease progression or unacceptable toxicities
Population: 20 participants were excluded because of ineligibility or absence in overall response evaluation.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | IMC-A12 | Temozolomide
Number analyzed (Participants) | 90 | 65
Proportion of Participants | 0.7667 [0.6793 to 0.8540] | 0.7846 [0.6847 to 0.8846]

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. Nine participants who were ineligible or did not receive treatment were excluded (both serious and other).
Groups:
- Group 1 (Chemotherapy, Radiation Therapy, Cixutumumab): Patients receive vincristine sulfate IV over 1 minute on day 1 of weeks 1-5, 7, 8, 11, 12, 15, 16, 20-24, 28, 29, 32, 33, 35, 38, 41-44, 47, 48, 50 & 51; irinotecan hydrochloride IV over 90 minutes on days 1-5 of weeks 1, 4, 20, 23, 47 & 50; ifosfamide IV over 1 hour and etoposide IV over 1-2 hours on days 1-5 of weeks 9, 13, 17, 26, & 30; doxorubicin hydrochloride IV over 1-15 minutes on days 1 and 2 of weeks 7, 11, 15, 28 & 32; cyclophosphamide IV over 30-60 minutes on day 1 of weeks 7, 11, 15, 28, 32, 35, 38, 41 & 44; dactinomycin IV over 1-5 minutes on day 1 of weeks 35, 38, 41 & 44; and cixutumumab IV over 1 hour on day 1 of weeks 1-51. Patients also undergo radiation therapy on days 1-5 of weeks 20-24.
  Cixutumumab: Given IV
  Cyclophosphamide: Given IV
  Dactinomycin: Given IV
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Irinotecan Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Vincristine Sulfate
Arm/Group | Group 1 (Chemotherapy, Radiation Therapy, Cixutumumab) | Group 2 (Chemotherapy, Radiation Therapy, Temozolomide)
Serious Adverse Events (participants affected / at risk) | 79/96 | 40/70
Other Adverse Events (participants affected / at risk) | 85/96 | 63/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Chemotherapy, Radiation Therapy, Cixutumumab) (N=96) | Group 2 (Chemotherapy, Radiation Therapy, Temozolomide) (N=70)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (10) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Death NOS (General disorders) | 30 (30) | 30 (30)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (12) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
GGT increased (Investigations) | 3 (4) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (10) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 6 (7) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 4 (6) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 3 (4) | 0 (0)
Lung infection (Infections and infestations) | 2 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (10) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5)
Neutrophil count decreased (Investigations) | 5 (9) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 8 (14) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 2 (2) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 8 (9) | 0 (0)
Serum amylase increased (Investigations) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 4 (8) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)
Weight loss (Investigations) | 6 (6) | 1 (1)
White blood cell decreased (Investigations) | 5 (10) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Chemotherapy, Radiation Therapy, Cixutumumab) (N=96) | Group 2 (Chemotherapy, Radiation Therapy, Temozolomide) (N=70)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 8 (10)
Acidosis (Metabolism and nutrition disorders) | 1 (3) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 15 (22) | 15 (22)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 9 (11) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 15 (18) | 12 (14)
Anxiety (Psychiatric disorders) | 5 (5) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 9 (12) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (7)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 7 (8) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 7 (10) | 9 (10)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Congenital, familial and genetic disorders - Other, specify (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (10) | 4 (4)
CPK increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 9 (9) | 3 (5)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 29 (32) | 12 (16)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Edema limbs (General disorders) | 3 (3) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 4 (4) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (2)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 35 (58) | 33 (56)
Fever (General disorders) | 6 (6) | 3 (3)
Fibrinogen decreased (Investigations) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GGT increased (Investigations) | 6 (9) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 4 (6)
Hematuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 20 (25) | 6 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 3 (4) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (7) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (7) | 5 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 13 (18) | 13 (17)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 11 (13) | 9 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (12) | 6 (8)
Hypotension (Vascular disorders) | 5 (6) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 15 (23) | 17 (22)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 2 (2) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 1 (1)
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 4 (4) | 4 (4)
Lung infection (Infections and infestations) | 1 (1) | 2 (2)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (5) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 9 (13) | 14 (17)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (13) | 7 (8)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (4) | 4 (4)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 21 (22) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 4 (5) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 2 (3)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 8 (10) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 3 (3) | 6 (6)
Serum amylase increased (Investigations) | 4 (5) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 2 (3) | 4 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Small intestine infection (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 6 (6)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 6 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (5) | 7 (9)
Urinary tract obstruction (Renal and urinary disorders) | 4 (5) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (11) | 9 (10)
Vulval infection (Infections and infestations) | 2 (2) | 0 (0)
Weight loss (Investigations) | 10 (13) | 2 (2)
White blood cell decreased (Investigations) | 6 (6) | 3 (5)
Wound infection (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less